CLINICAL TRIAL: NCT06934876
Title: Waveform Capnography and Colorimetric Carbon Dioxide Detection During Tracheal Intubation of Critically Ill Adults
Brief Title: Waveform Capnography Compared to Colorimetric Carbon Dioxide Detection During Tracheal Intubation of Critically Ill Adults
Acronym: WAVE
Status: Recruiting | Type: Observational
Sponsor: Brian Driver (Other)
Responsible Party: Sponsor-Investigator, Brian Driver, Co-Principal Investigator, Hennepin Healthcare Research Institute
Organization: Hennepin Healthcare Research Institute (Other)
Other Study IDs: IRB-FY2024-947
Record Dates: First submitted 2025-04-11; First posted 2025-04-18 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-10

CONDITIONS: Acute Respiratory Failure
Keywords: tracheal intubation; emergency intubation; waveform capnography; end-tidal CO2; exhaled carbon dioxide; colorimetric detection of exhaled carbon dioxide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Critically ill adults undergoing emergency tracheal intubation: Adult patients who are undergoing emergency intubation in the ED and ICU
  Interventions: Diagnostic Test: Colorimetric carbon dioxide (CO2) detection; Diagnostic Test: Waveform capnography

INTERVENTIONS:
Diagnostic Test: Colorimetric carbon dioxide (CO2) detection — All patients will undergo colorimetric carbon dioxide (CO2) detection. The reading will be assessed by a clinician at the bedside who will answer yes or no to the following question, asked after 7 breaths have been delivered following intubation: "Is the color change consistent with a tube located in the trachea?"
Diagnostic Test: Waveform capnography — All patients will undergo waveform capnography. The reading will be assessed by a clinician at the bedside who will answer yes or no to the following question, asked after 7 breaths have been delivered following intubation: " Is the waveform consistent with a tube located in the trachea?"

SUMMARY:
This study will compare the sensitivity and specificity of waveform capnography versus colorimetric carbon dioxide detection to identify tracheal placement of the endotracheal tube during intubation of critically ill adults.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is located in a participating unit (ED or ICU)
2. Patient is undergoing tracheal intubation.
3. The clinician intends to use an exhaled CO2 detection device to confirm tracheal placement of the tube.

Exclusion Criteria:

1. Patient is known to be a prisoner
2. Patient is known to be < 18 years old
3. A responsible clinician has determined that sole use of either waveform capnography or colorimetric testing is required for optimal care of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill adult patients undergoing emergency intubation
Sampling Method: Non-Probability Sample
Enrollment: 1332 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of the test of exhaled carbon dioxide to detect a endotracheal tube positioned in the trachea. | From intubation until 7 breaths from the ventilator are delivered, approximately 1 minute
  The co-primary endpoints are the sensitivity and speciﬁcity of each test (against the reference standard) to accurately detect the tube location.
  The sensitivity of each CO2 detection method describes the probability that the CO2 detection method is consistent with a tube location in the trachea for a patient who has an endotracheal tube located inside the trachea.
  The co-primary outcomes are a direct comparison of the sensitivity and specificity between the two index tests using McNemar's test with a two-sided P value with a significance level of 0.05. The McNemar's test is well-suited to paired data where both diagnostic tests are applied to the same patients. We will also present the absolute between-group difference with 95% confidence intervals.

SECONDARY OUTCOMES:
Specificity of the test of exhaled carbon dioxide to detect a endotracheal tube positioned outside of the trachea. | From intubation until 7 breaths from the ventilator are delivered, approximately 1 minute
  The co-primary endpoints are the sensitivity and specificity of each test (against the reference standard) to accurately detect the tube location. The specificity of each CO2 detection method describes the probability that the CO2 detection method is consistent with non-tracheal tube location for a patient who has an endotracheal tube located outside the trachea (e.g., esophageal intubation).
  The reference standard determines the tube location and will be categorized as trachea, non-tracheal, or indeterminate according to the approved protocol.
  The co-primary outcomes are a direct comparison of the sensitivity and specificity between the two index tests using McNemar's test with a two-sided P value with a significance level of 0.05. The McNemar's test is well-suited to paired data where both diagnostic tests are applied to the same patients. We will also present the absolute between-group difference with 95% confidence intervals.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Lahey Hospital & Medical Center, Burlington, Massachusetts
  - Hennepin Healthcare, Minneapolis, Minnesota
  - Duke University School of Medicine, Durham, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - The Ohio State University College of Medicine, Columbus, Ohio
  - Oregon Health and Sciences University, Portland, Oregon

IPD SHARING:
Plan to Share IPD: Yes
The authors will share the full de-identified dataset beginning 12 months after publication until 48 months after publication for researchers testing a hypothesis outlined in an institutional review board approved protocol. These data can be accessed by emailing the corresponding author. A signed data access agreement will be required.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: From 12 months after publication until 48 months after publication
Access Criteria: Researchers testing a hypothesis outlined in an institutional review board approved protocol can access the full de-identified dataset. These data can be accessed by emailing the corresponding author. A signed data access agreement will be required.